CLINICAL TRIAL: NCT04437329
Title: Nedaplatin Versus Cisplatin in Induction Chemotherapy Combined With Concurrent Chemoradiotherapy for Locally Advanced Nasopharyngeal Carcinoma：a Prospective, Parallel, Randomized, Open Labeled, Phase III Non-Inferiority Clinical Study
Brief Title: Nedaplatin Versus Cisplatin in Treatment for Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jin-Quan Liu, President of Affiliated Tumor Hospital of Guangzhou Medical University, Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPC-NDP
Record Dates: First submitted 2020-06-03; First posted 2020-06-18 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: induction chemotherapy; nedaplatin; cisplatin; concurrent chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Docetaxel; nedaplatin; Fluorouracil; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DNF-N (Experimental): 1. Induction chemotherapy:
     three cycles of intravenous docetaxel 60 mg/m² on day 1, intravenous nedaplatin 60 mg/m² on day 1, and continuous intravenous fluorouracil 600 mg/m² per day from day 1 to day 5, every 3 weeks
  2. Concurrent chemoradiotherapy:
     three cycles of 100 mg/m² nedaplatin every 3 weeks, concurrently with intensity-modulated radiotherapy
  3. Radiotherapy: radical intense modulated radiation therapy
  Interventions: Drug: Docetaxel, nedaplatin, fluorouracil; Drug: Nedaplatin; Radiation: Intensity modulated-radiotherapy
- DPF-P (Active Comparator): 1. Induction chemotherapy:
     three cycles of intravenous docetaxel 60 mg/m² on day 1, intravenous cisplatin 60 mg/m² on day 1, and continuous intravenous fluorouracil 600 mg/m² per day from day 1 to day 5, every 3 weeks
  2. Concurrent chemoradiotherapy:
     three cycles of 100 mg/m² cisplatin every 3 weeks, concurrently with intensity-modulated radiotherapy
  3. Radiotherapy: radical intense modulated radiation therapy
  Interventions: Drug: Docetaxel, cisplatin, fluorouracil; Drug: Cisplatin; Radiation: Intensity modulated-radiotherapy

INTERVENTIONS:
Drug: Docetaxel, nedaplatin, fluorouracil — Induction chemotherapy. Docetaxel 60 mg/m2 intravenous day1. Nedaplatin 60 mg/m2 intravenous day1. Fluorouracil 3000 mg/m2 continuous intravenous infusion 120 hours from day1. Every 21 days, 3 cycles.
  Other Names: DNF
  Arms: DNF-N
Drug: Docetaxel, cisplatin, fluorouracil — Induction chemotherapy. Docetaxel 60 mg/m2 intravenous day1. Cisplatin 60 mg/m2 intravenous day1. Fluorouracil 3000 mg/m2 continuous intravenous infusion 120 hours from day1. Every 21 days, 3 cycles.
  Other Names: DPF
  Arms: DPF-P
Drug: Nedaplatin — Concurrent chemotherapy. Nedaplatin 100 mg/m2 intravenous at day1, 22, 43 of radiotherapy.
  Other Names: NDP
  Arms: DNF-N
Drug: Cisplatin — Concurrent chemotherapy. Cisplatin 100 mg/m2 intravenous at day1, 22, 43 of radiotherapy.
  Other Names: DDP
  Arms: DPF-P
Radiation: Intensity modulated-radiotherapy — Intensity modulated-radiotherapy (IMRT) is given as 2.0-2.33 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 66 Gy or greater to the primary tumor.
  Other Names: IMRT

SUMMARY:
To compare the effectiveness and toxicity of nedaplatin versus cisplatin in induction chemotherapy combined with concurrent chemoradiotherapy for locoregionally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
This is a prospective, parallel, randomized, open labeled, phase III, non-inferiority clinical trial to compare the effectiveness and toxicity of nedaplatin versus cisplatin in induction chemotherapy combined with concurrent chemoradiotherapy for locoregionally advanced nasopharyngeal carcinoma patients in endemic area - nedaplatin, docetaxel and fluorouracil as induction chemotherapy regimen combined with nedaplatin as concurrent chemoradiotherapy (DNF-N) versus cisplatin, docetaxel and fluorouracil as induction chemotherapy regimen combined with cisplatin as concurrent chemoradiotherapy (DPF-P). All patients will receive radical intense modulate radiation therapy (IMRT). The primary endpoint is progress free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, including WHO II or III
2. Original clinical staged as III-IVa (except T3-4N0) according to the 8th edition American Joint Committee on Cancer staging system
3. No evidence of distant metastasis (M0)
4. Age between 18-65
5. WBC≥4×10^9/ l, platelet ≥ 100×10^9/ l and hemoglobin ≥ 90g/l
6. With normal liver function test (TBIL、ALT、AST ≤ 2.5×uln)
7. With normal renal function test (creatinine ≤ 1.5×uln or ccr ≥ 60ml/min)
8. Satisfactory performance status: KARNOFSKY scale (KPS) > 70
9. Patients must give signed informed consent

Exclusion Criteria:

1. Histologically confirmed keratinizing nasopharyngeal carcinoma (WHO I)
2. Age >65 or < 18 years
3. Treatment with palliative intent
4. Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer
5. History of previous radiotherapy, chemotherapy, or surgery (except diagnostic) to the primary tumor or nodes
6. History of previous radiotherapy
7. Pregnancy or lactation
8. Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, acute exacerbation of chronic obstructive pulmonary disease or other respiratory illness requiring admission to hospital, active hepatitis, and mental disturbance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Progress-Free Survival (PFS) | 3 years
  Progress-free survival is calculated from the date of randomisation to the date of locoregional failure, distant failure, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival(OS) | 3 years
  The OS was defined as the duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up.
Locoregional Relapse-Free Survival(LRRFS) | 3 years
  Relapse-free survival was defined as the time from random assignment to local or regional relapse, or death from any cause.
Distant metastasis-Free Survival(DMFS) | 3 years
  Distant metastasis-free survival was defined as the time from random assignment to distant metastasis, or death from any cause.
Quality of life (QoL) | 3 years
  Quality of life (QoL) was assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire module for head and neck (EORTC QLQ-H&N35). The EORTC QLQ-H&N35 scale employs a 4-point response format ("not at all" to "very much"). Scale scores are transformed to a scale from 0 to 100 according to the EORTC scoring algorithm. For the functioning and the global QoL scale, a higher score indicates better health. For the symptom scales, a higher score indicates a higher level of symptom burden. Either English or Chinese version will be used according to patient's language habits.
Objective Response Rate (ORR) | 12 weeks after the interventions
  Objective Response Rate (ORR) were assessed with nasopharyngeal and neck MRI and flexible nasopharyngoscopy, according to the Response Evaluation Criteria in Solid tumors(version 1.1)
Disease Control Rate (DCR) | 12 weeks after the interventions
  Disease Control Rate (DCR) were assessed with nasopharyngeal and neck MRI and flexible nasopharyngoscopy, according to the Response Evaluation Criteria in Solid tumors(version 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Jinquan Liu, M.D, Study Director — Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Locations (1):
- Department of radiotherapy(Section 5),Affiliated Cancer Hospital & Institute of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No